CLINICAL TRIAL: NCT01439737
Title: Metabolomic Analysis of Exhaled Breath Condensate, Plasma and Urine Specimens in Adult Asthmatics
Brief Title: Metabolomic Analysis of Exhaled Breath Condensate in Asthmatics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201108051RC
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Asthma
Keywords: Asthma; metabolomics; exhaled breath condensate
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled breath condensates, serum, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- asthma

SUMMARY:
Asthma is a chronic inflammatory airway disease. Significant heterogeneity exists in the clinical manifestations and treatment responses in these patients. Metabolomics is a large-scale approach to monitoring as many as possible of the compounds involved in cellular processes in a single assay to derive metabolic profiles. Compared with genomics or proteomics, metabolomics reflects changes in phenotype and therefore function. Up to now, few studies have evaluated the role of metabolomic analysis in the diagnosis and prognostic evaluation of airway disorders. Collection of exhaled breath condensate (EBC) is a newly developed, noninvasive method that may allow clinicians and researchers to assess biochemical profiles in the alveolar lining fluid. This study will apply metabolomics to examine the biomarkers in the EBCs, serum and urine specimens in adult asthmatics.

DETAILED DESCRIPTION:
The aims of this study are: 1. Metabolomic profiling of the exhaled breath condensate (EBC), serum and urine specimens in adult asthmatics; 2. Correlation between metabolomic profiles of these specimens with the severity and control of asthma; 3. Comparing metabolomic profiles in asthmatics with different phenotypes and endotypes; 4.Comparing metabolomic profiles obtained from asthmatics during stable and acute exacerbation periods; 5. Comparing metabolomic profiles in asthmatics before and after inhaled corticosteroid therapy.

ELIGIBILITY:
Inclusion Criteria:

1. 20-90 years
2. Diagnosis of asthma based on the GINA guideline

Exclusion Criteria:

1. Patient with cancer
2. Patient with long-term ventilator use

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult asthmatics
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Hung Kuo, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Internal Medicine, National Taiwan University Hospital, Taipei, Taiwan